CLINICAL TRIAL: NCT01603498
Title: Preemptive Effect of Dexamethasone and Methylprednisolone on Pain, Swelling and Trismus After Third Molar Surgery: a Split-mouth Randomized Triple-blind Clinical Trial
Brief Title: Effect of Dexamethasone and Methylprednisolone on Pain, Swelling and Trismus After Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 053/10
Record Dates: First submitted 2012-05-17; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Pain,; Edema,; Trismus
Keywords: pain measurement,; edema,; trismus
MeSH Terms: conditions — Pain; Edema; Trismus | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone 8mg (Experimental)
  Interventions: Drug: Dexamethasone
- Methylprednisolone (Experimental): Methylprednisolone 40mg
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 8mg
  Other Names: Dexametasone acetate
  Arms: Dexamethasone 8mg
Drug: Methylprednisolone — Methylprednisolone 40mg
  Arms: Methylprednisolone

SUMMARY:
The main aim of the present study was to investigate the effect of preemptive dexamethasone and methylprednisolone to prevent pain, swelling and limitation in mouth opening following third molar extraction.

DETAILED DESCRIPTION:
Third molar surgery is often associated with significant post-surgical sequelae. The trauma caused to soft and bony tissue can result in considerable pain, swelling and trismus. Symptoms begin gradually having a peak 2 days after extraction. The use of corticosteroids such as dexamethasone and methylprednisolone can be a valuable tool when performing moderate to moderately severe oral surgical procedures. No clear consensus have emerged yet regarding patient selection, dosage, timing and type of administration of steroid. In this light, this clinical trial aim to compare the effect of preemptive dexamethasone and methylprednisolone to prevent pain, swelling and limitation in mouth opening following third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of asymptomatic bilateral extractions of lower third molars
* Aged 18 years or older;
* Have a good health and no disease;

Exclusion Criteria:

* Patients with history of any medication treatment within 15 days before the beginning of the research, history of allergy to the drugs, substances or materials used in this study, pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative sequelae following thir molar extraction | up to seven days postoperative
  During the postoperative intervals of 24, 48 and 72 hours and seven days, the swelling was determined using linear measures in the face and trismus by maximum mouth opening. The postoperative pain was self-recorded by the patient using visual analogue scale in 72 hours with an interval of eight hours

SECONDARY OUTCOMES:
Analgesic consumption; duration of surgery | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Eduardo Alcântara, MsC, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil